CLINICAL TRIAL: NCT02307539
Title: Feasibility of an Interdisciplinary Palliative Care Planning Intervention in Pancreatic Cancer
Brief Title: Palliative Care in Improving Quality of Life in Patients With Newly Diagnosed Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14273; NCI-2014-02367 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14273 (Other: City of Hope Medical Center); U24NR014637 (NIH)
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Stage IIA Pancreatic Cancer; Stage IIB Pancreatic Cancer; Stage III Pancreatic Cancer; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Psychiatric Rehabilitation; Palliative Care; Patient Comfort

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (PCPI intervention) (Experimental): Patients receive a handbook titled "Supporting You During Cancer Treatment" with educational material on QOL issues. Patients undergo 2 education sessions on handbook material in-person or by telephone, with session 1 focusing on physical and social well-being issues and session 2 focusing on psychological and spiritual well-being issues. At the beginning of each session, patients select 3 priority topics from a list, and content is tailored to patient needs.
  Interventions: Procedure: Psychosocial Assessment and Care; Other: Palliative Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Psychosocial Assessment and Care — Undergo PCPI
  Other Names: Psychosocial Assessment; Psychosocial Care; Psychosocial Care/Assessment; Psychosocial Studies; Psychosocial Support
Other: Palliative Therapy — Undergo PCPI
  Other Names: Comfort Care; Palliative Care; Palliative Treatment; Symptom Management
Other: Quality-of-Life Assessment — Undergo QOL assessment
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Undergo questionnaire administration

SUMMARY:
This pilot clinical trial studies a palliative care program in improving the quality of life of patients with newly diagnosed pancreatic cancer. Palliative care is care given to patients who have a serious or life-threatening disease, and focuses on managing disease symptoms, side effects of treatment or the disease, and improving patient quality of life. Studying a palliative care program used for other types of cancer may help doctors learn whether it can improve the quality of life of patients with pancreatic cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To pilot-test an interdisciplinary Palliative Care Planning Intervention (PCPI) in pancreatic cancer. Specifically, to describe patients' satisfaction with the timing, content, and delivery of the PCPI intervention.

SECONDARY OBJECTIVES:

I. To pilot-test all selected measures for the study, including measures for healthcare resource utilization, overall cost, and patient/family out of pocket expenses.

II. The long-term objective of this pilot study is to conduct a larger PCPI intervention study for pancreatic cancer patients and evaluate its impact on quality of life (QOL), symptom intensity, healthcare resource utilization, and healthcare costs.

OUTLINE:

Patients receive a handbook titled "Supporting You During Cancer Treatment" with educational material on QOL issues. Patients undergo 2 education sessions on handbook material in-person or by telephone, with session 1 focusing on physical and social well-being issues and session 2 focusing on psychological and spiritual well-being issues. At the beginning of each session, patients select 3 priority topics from a list, and content is tailored to patient needs.

After completion of study, patients are followed up at 1 and 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed, new diagnosis of borderline resectable, locally advanced resectable/unresectable, or metastatic pancreatic cancer
* Patients who are scheduled to receive treatments (neoadjuvant therapy, surgery, adjuvant therapy, or palliative chemotherapy) at City of Hope (COH)
* All subjects must have the ability to understand and the willingness to provide informed consent

Exclusion Criteria:

* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-11; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Reasons for refusal to participate | Up to 2 months
  Descriptive statistics will be provided.
Reasons for failure to complete study | Up to 2 months
  Descriptive statistics will be provided.
Attendance at two educational sessions | Up to 2 months
  Descriptive statistics will be provided.
Completion of intervention | Up to 2 months
  Descriptive statistics will be provided.
Patient satisfaction with timing, content, and delivery of PCPI | Up to 2 months
  Presented through summary statistics of data from the patient satisfaction tool.
Qualitative interview data | Up to 2 months
  Each interview transcript will be initially reviewed to provide a glimpse of potential domains and targets. Content analysis will be conducted on the transcribed qualitative data. Transcripts will be assigned codes. Content analysis occurring through coding consisting of line-by-line analysis with themes identified will be initiated. The research team will independently analyze selected segments of the data to verify themes. Coding will be checked and validated by the principal investigator and research team.

SECONDARY OUTCOMES:
Healthcare resource utilization, as measured by the Report of Healthcare Services Form | Up to 2 months
  Data will be summarized using descriptive statistics. Established instruments will be scored according to standard instructions, and appropriate descriptive statistics computed.
Overall cost, as measured by the Finances and Out of Pocket Costs Tool | Up to 2 months
  Data will be summarized using descriptive statistics. Established instruments will be scored according to standard instructions, and appropriate descriptive statistics computed.
Patient/family out of pocket expenses, as measured by the Finances and Out of Pocket Costs Tool | Up to 2 months
  Data will be summarized using descriptive statistics. Established instruments will be scored according to standard instructions, and appropriate descriptive statistics computed.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States